CLINICAL TRIAL: NCT06183294
Title: Evaluation of a Novel Non-Invasive Automated Fractional Flow Reserve Software System in Patients With Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: MedHub-AI (Unknown)
Responsible Party: Principal Investigator, Ehtisham Mahmud, Professor and Division Chief, Cardiovascular Medicine, University of California, San Diego
Other Study IDs: 808066
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Stable Angina, Unstable Angina, NSTEMI
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- : adult subjects who underwent a clinically indicated invasive coronary angiography: adult subjects with stable angina, unstable angina or NSTEM1 who underwent a clinically indicated invasive coronary angiography and on whom invasive FFR has been measured in vessels with coronary lesions.
  Interventions:
  Other: Collecting invasive FFR measurements.
  Interventions: Other: Collecting invasive FFR measurements.

INTERVENTIONS:
Other: Collecting invasive FFR measurements. — Invasive FFR measurements from the patient's hospital records will be collected.
  Other Names: Data collection

SUMMARY:
This retrospective study will evaluate the coronary angiograms of approximately 100 patients who have undergone invasive angiography and fractional flow reserve (FFR). DICOM files of the angiograms will be analyzed on a secure computer within the cardiac catheterization laboratory using the AutocathFFR software to assess if invasive FFR measurements and automated computer analysis of FFR measurements correlate. AutocathFFR measurement per lesion will be compared to the gold standard, invasive FFR value, where an FFR ≤ 0.80 will be considered "positive", while an FFR > 0.8 will be considered "negative". The AutocathFFR value will be compared to the invasive FFR measurements. The sensitivity and specificity of the AutocathFFR will be calculated, as well as the AutocathFFR accuracy, positive predictive value and negative predictive value per lesion. Device success will be calculated as the ratio of completed versus initiated AutocathFFR index calculations. Usability of the AutocathFFR software will be evaluated using dedicated questionnaires to be completed by the user (cardiologists).

DETAILED DESCRIPTION:
Coronary angiography is the gold standard for assessment of coronary artery disease. Coronary artery stenosis in lesions in the mild and severe range are easily interpreted by clinicians as meeting thresholds for clinical and hemodynamic significance. Moderate coronary artery disease remains an area of investigation and assessment as lesions in the 50-70% range are often unclear in their hemodynamic and clinical significance. Indices of coronary perfusion such as fractional flow reserve (FFR) have been developed to assess whether lesions are hemodynamically significant and could potentially benefit from revascularization. Assessment of FFR however requires further invasive testing, manipulation, and equipment, each with risk to the patient. We aim to retrospectively assess a non-invasive FFR software, the AutocathFFR system in the evaluation of coronary artery disease in patients who underwent invasive measurements to assess the accuracy of this system.

This study will assess the performance (sensitivity, specificity, accuracy) of the AutocathFFR measurements obtained from angiograms for the non-invasive determination of the presence of hemodynamically significant coronary lesions. The software device will be run on angiograms generated during cardiac catheterization and will be compared to the gold standard, invasive fractional flow reserve (FFR) measurements.Invasive coronary angiography (ICA) has long been considered the reference standard technique for the diagnosis of coronary artery disease (CAD). Decisions regarding revascularization procedures have traditionally been based on the visual assessment of coronary stenosis severity. However, this strategy is being challenged based on increasing recognition of the limitations of visual interpretation of conventional angiographic images. One of the major concerns is considerable inter-observer variability in interpretation of coronary angiograms1. Even the use of quantitative techniques has not substantially improved the predictive value of ICA for identifying the presence of lesion-specific ischemia2. Even more importantly, it is now recognized that many additional factors may collectively influence flow dynamics in a vessel in addition to the degree of narrowing at any single point. Accordingly, current evidence and guidelines stipulate that the decision to proceed to revascularization should be governed by the hemodynamic significance of a lesion, rather than angiographic severity alone, particularly for borderline ("gray zone") lesions. Currently, measurement of Fractional Flow Reserve (FFR) is the preferred technique for invasive assessment of flow limitation.

Fractional Flow Reserve, or FFR, is a measure usually gauged by an invasive wire that can accurately measure blood pressure in a specific part of the coronary artery. The wire is inserted through a standard diagnostic catheter at the time of a coronary angiogram and measurements obtained during hyperemic stimulus, typically with the use of intravenous or intracoronary adenosine.

An FFR value equal or less than 0.8 is generally considered to be the best discriminator of flow obstruction and the most relevant predictor of improved clinical outcome after coronary revascularization3,4. Trials such as Fractional Flow Reserve versus Angiography for Guiding Percutaneous Coronary Intervention (FAME) 5,6, whereas those without ischemia receive little benefit, or even harm, with revascularization. Further, the Deferral Versus Performance of Percutaneous Coronary Intervention of Non-Ischemia-Producing Stenoses, (DEFER) trial has shown that patients with non-flow-limiting lesions do not require intervention and show favorable outcomes with use of optimal medical therapy alone, with annual rates of myocardial infarction and mortality of less than 1%7. Accordingly, evaluation of the hemodynamic significance of coronary stenosis during ICA by using pressure wire-derived FFR, an approach that allows combined anatomic and physiologic assessment, has become a cornerstone to determine lesion-specific ischemia and appropriate decision making8,9. Furthermore based on the above studies, the American (ACC/AATS/AHA/ASE/ASNC/SCAI/SCCT/ STS 2017 Appropriate Use Criteria for Coronary Revascularization in Patients with Stable Ischemic Heart Disease10) and European (ESC/EACTS Guidelines on myocardial revascularization11) Guidelines recommend the routine use of FFR for further defining the need for revascularization.

Nevertheless, there are several risks associated with invasive FFR, including the use of an invasive pressure wire through the coronary arteries, drift in the pressure wire reading, side effects from hyperemic agents, the additional time required to perform the procedure in multiple blood vessels, as well as other technical challenges associated with the procedure. For these reasons, as well as others, such as costs and time, invasive FFR is not employed in many procedures even though it may provide clinically useful information.

As physiology-guided revascularization is important as pointed out by the American and European Guidelines, non-invasive techniques for measuring FFR have been developed. The ability to simulate the value measured by invasive FFR devices by computer models has been demonstrated by several devices.

ELIGIBILITY:
Inclusion Criteria:

* patients who are >18 years of age, undergone a coronary angiogram for a clinically indicated reason, and who underwent coronary hemodynamic testing with invasive FFR.

Exclusion Criteria:

* Invasive FFR not obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of coronary angiograms of 100 consecutive patients who have undergone fractional flow reserve (FFR) testing within our institution
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
To assess the performance (sensitivity, specificity, accuracy) of the AutocathFFR measurements obtained from angiograms for the non-invasive determination of the presence of hemodynamically significant coronary lesions. | 2 months
  The software device will be run on angiograms generated during cardiac catheterization and will be compared to the gold standard, invasive fractional flow reserve (FFR) measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Ehtisham Mahmud, MD, Principal Investigator — UC San Diego Health
Locations (1):
- UC San Diego Health, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No